CLINICAL TRIAL: NCT04124666
Title: Clinical Study of Allogeneic Granulocyte Infusion in the Treatment of Patients With Advanced Cancer
Brief Title: Clinical Study of Granulocyte Infusion for Advanced Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2019-01
Record Dates: First submitted 2019-09-10; First posted 2019-10-11 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Granulocytes infusion only (Experimental): Fresh, non-irradiated granulocytes from ABO, Rh, CMV compatible, unrelated donors; bioactivity of anti-cancer ability meets the criteria.
  Interventions: Biological: Granulocytes

INTERVENTIONS:
Biological: Granulocytes — Granulocytes cross-matched for ABO-Rh and CMV; bioactivity of anti-cancer ability meets the criteria.

SUMMARY:
Background & Rationale:

For years, most tumor immunotherapy researches have focused on T cell and natural killer (NK) cell therapies, most of which involve amplification and modification of the patient's immune cells for reinfusion therapy. However, for the treatment of solid tumors, there is currently little breakthrough. Recently, researchers have reported a colony of cancer-resistant mice developed from a single mouse that was immune to multiple lethal cancer cell injections. Further research revealed that such anti-cancer immunity can cause rapid shrinkage or disappearance of the tumors in other cancer-bearing mice. Interestingly, this therapeutic effect is due to the donor granulocytes, instead of T cells or NK cells. Infusion of granulocytes is a classic therapy in treating infection associated with granulocytopenia. Currently, clinical collection of blood components, including isolation of granulocytes, is a mature technique. The infusion of granulocytes is a viable anticancer therapy combining the classic technique and novel anticancer approach. This proposed trial will test whether granulocyte infusions from healthy unrelated donors can be used to treat advanced cancer. In the proposed trial, up to 100 Subjects with advanced cancer can be entered. Each patient will be given a dose of (2.0-5.0)x10^10 granulocytes from a different healthy donor every week over a course of 5 doses. The trial will evaluate the subject's cancer 7, 30, 90 and 180 days after the last infusion.

DETAILED DESCRIPTION:
Granulocyte anti-cancer therapy refers to a method in which healthy donor granulocytes with high cancer-killing activity are collected and infused into a specific cancer patient by matching, to achieve the therapeutic anticancer effect. In this proposed trial, up to 100 Subjects with advanced cancer can be entered. Potentially hundreds of healthy Donor-participants will be recruited. First, granulocyte donors will be identified via in-vitro assay of Cancer Killing Activity (CKA), which screens healthy Donor-participants for those with anticancer activity of more than 80%. Secondly, after donor-recipient blood matching, (2.0-5.0)x10^10 granulocytes will be collected from each donor, accounting for about 1/10 of the human body. Each patient will be given a dose of (2.0-5.0)x10^10 granulocytes from a different donor per week over a course of 5 doses (with an ideal total infusion of 2X10^11 granulocytes). After each infusion, the patients will be monitored carefully for possible adverse events. If adverse events occur, the infusion can be slowed down or stopped until the adverse events can be managed. The trial will observe the subject's cancer 7, 30, 90 and 180 days after the last infusion. Target lesions, non-target lesions, and new lesions will be evaluated via medical imaging and tumor markers. The responses will be compared against the measurements at baseline.

ELIGIBILITY:
Inclusion Criteria for Subjects:

* Malignant tumor confirmed by puncture pathology/postoperative pathology;
* Clinical stage IV;
* Performance status of ≤2 on the ECOG scale
* Life expectancy of at least 3 months
* All patients was diagnosed metastatic tumor by histology and cytology. Cytoreductive surgery can be performed if the patient can endure surgery.
* Measurable Disease: Lesions that can be accurately measured in at least one dimension (longest diameter recorded) as 20 mm with conventional technique or as 10 mm with spiral CT scan.If the lesion is between 15mm and 20mm, the thickness of the CT layer should be no more than 0.5mm. For multiple lesions, select a representative 10 lesions (maximum 5 in the same organ) and calculate the sum of the longest diameters of all target lesions as the baseline sum diameter.
* ≥ 4 weeks since prior medical therapy, radiation therapy, and surgery
* Laboratory tests meet the following criteria:

A. Bone marrow function: Absolute blood neutrophil (ANC) count ≥1*10^9 /L, blood small (PLT) ≥75*10^9 /L.

B. Liver function: serum total bilirubin (STB), combined bilirubin (CB) ≤ upper limit of normal (ULN) * 1.5, alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ULN*2.5 (in the absence of liver metastases), or ≤ULN*5 (with liver metastases);

C. Renal function: serum creatinine (Cr) ≤ ULN * 1.5, endogenous creatinine clearance (Ccr) ≥ 50 mL / min (calculated using the Cockcroft-Gault formula, see Appendix 2);

* The anti-neutrophil antibody test result was negative.
* The patient volunteered and signed an informed consent form.

Exclusion Criteria of Subjects:

* Arrhythmia, congestive heart failure, or severe coronary artery disease;
* Pregnant or nursing women;
* Patients with severe autoimmune diseases;
* Patients who have been using or are using immunosuppressive agents for a long time;
* Those with coagulopathy;
* Cases that the investigator considered inappropriate for inclusion.

Inclusion Criteria for Granulocyte Donors:

* Must have signed Donor-participant Informed Consent Form
* Must be able to provide granulocytes in local blood donation center, and transport collected granulocytes to the hospital blood bank or clinical application within 24 hours;
* Must score >80% in Cancer Killing Assay (CKA), a score of 60-80% would be considered when there are insufficient donors;
* Must have CMV negative or positive sero-testing completed; only seronegative donors are accepted for a seronegative recipient;
* Must have compatible ABO and RH typing with the recipient;
* Must be qualified for blood donation: aged 18-35, male >50kg or female >45kg, normal cardiopulmonary function, specific gravity of blood male≥1.052 or female≥1.051, HbsAg, anti-HCV, anti-HIV, or syphilis tests.

Exclusion Criteria for Granulocyte Donors:

* Dental or other minor surgery within preceding 15 days;
* Arrhythmia, congestive heart failure, or severe coronary artery disease;
* Major surgery within preceding 6 months;
* Appendectomy, hernia repair, or tonsillectomy within preceding 3 months;
* Females 3 days before or after menstruation, ≤6 months since prior pregnancy or abortion, ≤ 1 year since delivery/breastfeeding;
* Recovery from flu or acute gastroenteritis within preceding week, acute renal infection within preceding month, pneumonia within preceding 3 months;
* Recovery from infectious diseases such as dysentery within preceding 6 months, typhoid fever within preceding year, brucellosis within preceding 2 years, or malaria within preceding 3 years;
* Recovery from localized dermatitis within preceding week, extensive inflammation within preceding 2 weeks;
* Receiving whole blood or blood components within preceding 5 years;
* Allergic to G-CSF mobilizer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 90 days post treatment
  The trial will observe the subject's progression free survival for 3 months after the granulocyte infusions are completed.

SECONDARY OUTCOMES:
median Overall Survival (mOS) | 180 days post treatment
  The patients will be followed 1 week, 1 month, 3 months and 6 months after the last treatment. Median Overall Survival will be measured as the length of time from the date of inclusion that half of the patients are still alive.
Objective Response Rate (ORR ) | 180 days post treatment
  Objective Response Rate will be evaluated based on the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. If a response is achieved in a patient, the evaluation will be repeated 4-6 weeks after the first evaluation to confirm the response.
Disease Control Rate (DCR) | 180 days post treatment
  Disease Control Rate will be measured as the percentage of patients achieved complete response (CR), partial response (PR) and stable disease (SD) to the treatment (evaluated based on RECIST 1.1).
Quality of life measured in ECOG | 180 days post treatment
  ECOG Scale of Performance Status will be evaluated for patients after treatment to reflect impact on quality of life.
Treatment-related adverse events | 5 weeks of treatment and 1 month post treatment
  Incidence of treatment-related adverse events as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongming Liu, MD/Ph.D, Principal Investigator — Shanghai East Hospital, Shanghai Tongji University
Locations (1):
- Department of Oncology, Shanghai East Hospital, Shanghai, Shanghai Municipality, China